CLINICAL TRIAL: NCT02403765
Title: Realization of Diagnostic Tools for the Early Analysis of Parkinson's Disease Through the Identification of Genetic Risk Profiles
Brief Title: Diagnostic Tools for Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Antonio Simeone, Head, Neuromed IRCCS
Other Study IDs: SMN01
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples for DNA extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Family cases: Family-based Parkinson patients carrying genetic variants associated with the disease
- Family controls: Family-based Control subjects

SUMMARY:
The study aims to identify genetic variants associated to Parkinson's disease through the analysis of exome-sequencing data of familial cases and controls. The identified variants will be used to generate a diagnostic tool for the identification of genetic risk profiles.

DETAILED DESCRIPTION:
1. Clinical evaluation of PD patients and relatives
2. High throughput analysis of genetic variants in genome exomes
3. Genotype-phenotype association testing
4. Identification of genetic risk variants for PD

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two out the following cardinal signs: resting tremor, cogwheel rigidity, bradykinesia, asymmetrical onset of symptoms and symptomatic response to L-dopa (levodopa)

Exclusion Criteria:

* Previous thalamotomy on the implanted sided, significant brain atrophy or structural damage seen on CT or MRI, marked cognitive dysfunction, active psychiatric symptoms, or concurrent neurological or other uncontrolled medical disorders.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the Center for Parkinson's disease of the IRCCS Neuromed, according to specific inclusion criteria. Approximatey 500 subjects, 30 years of age or older, recruited with a family-based approach, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Identification of genetic variants associated with Parkinson's disease | Two years
  Analysis of exome sequencing data; annotation of genetic variants; selection of variants present in cases and absent in controls

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simeone, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy